CLINICAL TRIAL: NCT02974088
Title: A Randomised, Assessor Blinded "Proof of Concept" (Phase IIa) Clinical Study to Assess the Efficacy and Safety of Nice 'n Clear Head Lice Lotion in the Treatment of Head Lice
Brief Title: Neem Lotion With Combing for Lice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Entomology Centre (Industry)
Collaborators: Leeds Health Protection Unit (Unknown); PN Lee Statistics and Computing Ltd (Unknown); Nelsons (Other)
Responsible Party: Principal Investigator, Ian F Burgess, Director, Medical Entomology Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTNC01
Record Dates: First submitted 2016-11-21; First posted 2016-11-28 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pediculoses; Head Lice
MeSH Terms: conditions — Lice Infestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neem-based lotion plus louse comb (Experimental): Neem-based conditioning lotion plus head louse detection and removal comb
  Interventions: Device: Neem-based lotion plus louse comb
- Neem-based lotion plus grooming comb (Experimental): Neem-based conditioning lotion plus regular grooming comb
  Interventions: Device: Neem-based lotion plus grooming comb

INTERVENTIONS:
Device: Neem-based lotion plus louse comb — Neem-based conditioning lotion was applied to washed and towel dried hair followed by systematic combing using a head louse detection and removal comb
  Other Names: Nice 'n Clear
  Arms: Neem-based lotion plus louse comb
Device: Neem-based lotion plus grooming comb — Neem-based conditioning lotion was applied to washed and towel dried hair followed by combing through using a regular grooming comb
  Other Names: Nice 'n Clear
  Arms: Neem-based lotion plus grooming comb

SUMMARY:
This was a Phase IIa randomised, assessor blinded, parallel group study in which half the participants were treated with Nice 'n Clear neem-based conditioning lotion plus combing with a head louse detection and removal comb and the remainder were treated with Nice 'n Clear plus combing with a normal grooming comb

DETAILED DESCRIPTION:
Neem oil has had a long reputation for killing a wide range of insects, including head lice. Several products are marketed with this oil as a named active ingredient, e.g. Nice 'n Clear neem-based conditioning lotion. This product was developed as an aid to combing out head lice for eliminating infestation but it has been considered possible that the neem oil could act to kill lice and inhibit their eggs from hatching.

This study was designed to compare use of Nice 'n Clear neem-based conditioning lotion when used with two different types of comb. One arm of the study was planned so that participants were combed using a plastic louse detection and removal comb (wet combing with conditioner method), in which it was expected the combing process would play a major role in efficacy. The other arm was planned so that participants were combed using a regular grooming comb, which would normally have little effect for removing head lice from the hair.

Comparison of the efficacy outcome in the two groups would determine whether the Nice 'n Clear neem-based conditioning lotion exhibited any effect to eliminate infestation independent of the combing

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are found to have an active head louse infection, i.e. the presence of live lice. Detection combing will be done with a fine-toothed plastic detection comb, until at least one louse is found.
* People who give written informed consent and/or, if the participant is below 16 years of age, whose guardian gives written informed consent to participate in the study. Assent/verbal assent forms will be required for those between the ages of 4 and 16 years of age. There is no maximum age limit.
* Participants must be available for the duration of the study i.e. 15 days.

Exclusion Criteria:

* People who have been treated with other head louse products within the previous 2 weeks (14 days).
* People who have undergone a course of antibiotic treatment using Cotrimoxazole, Trimethoprim or Septrin within the previous 4 weeks, or who are currently taking such a course.
* People whose hair has been bleached, colour treated, or semi-permanently waved within the previous 2 weeks, this includes the use of semi-permanent colouring agents. Home use wash in/wash out colouring agents are acceptable.
* People who have taken part in another clinical study within 4 weeks prior to entry to this one.
* Females who are pregnant or breast-feeding.
* Participants who have already taken part in this study.
* People who have a known allergy to any of the ingredients of Nice 'n Clear Lotion (including allergy to Paraben preservatives)
* Children under 6 months of age.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian F Burgess, Principal Investigator — Medical Entomology Centre
Locations (1):
- Medical Entomology Centre, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Contact Principal Investigator

REFERENCES:
- See also: Final Report Summary - ClearBrush (A Novel Integrated Ultrasonic Brush and Sonically Activated Lotion to Provide a Full System Approach to the Eradication of the European Head Louse Menace) — http://cordis.europa.eu/result/rcn/46970_en.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment between 26 May 2006 and 31 August 2006. Community recruitment with domiciliary visits
Pre-assignment Details: None defined
Period: Overall Study
Arm/Group | Neem-based Lotion Plus Louse Comb | Neem-based Lotion Plus Grooming Comb
Started | 23 | 24
Completed | 23 | 21 (Nurse left without notice and took CRFs and data for 2 subjects.)
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neem-based Lotion Plus Louse Comb | Neem-based Lotion Plus Grooming Comb | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 19 | 39
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Head Louse Infestation as Assessed by Detection Combing
Description: Recruitment at Day 0. Success of treatment = No lice present at Day 14 and no lice present at Day 10
Time Frame: 15 days
Population: All participants who completed the 15 study days
Measure: Count of Participants; unit: Participants
Arm/Group | Neem-based Lotion Plus Louse Comb | Neem-based Lotion Plus Grooming Comb
Number analyzed (Participants) | 23 | 22
Participants | 23 | 22

2. Secondary Outcome: Difference in Number of Participants Free From Head Louse Infestation According to Comb Type Used
Description: It was expected that the louse comb group would show a high level of success (elimination of infestation). The measure of efficacy of the neem-based lotion was the relative efficacy observed in the grooming comb group compared with the louse comb group
Time Frame: 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Neem-based Lotion Plus Louse Comb | Neem-based Lotion Plus Grooming Comb
Number analyzed (Participants) | 23 | 24
Participants | 23 | 22

3. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Number of participants with application site reactions such as irritation, erythema, or other events related to treatment
Time Frame: 15 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Neem-based Lotion Plus Louse Comb | Neem-based Lotion Plus Grooming Comb
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 1/23 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neem-based Lotion Plus Louse Comb (N=23) | Neem-based Lotion Plus Grooming Comb (N=24)
Application site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No